CLINICAL TRIAL: NCT03063463
Title: Mechanisms of Weight Loss in Patients Diagnosed With Achalasia: A Prospective Observational Study
Brief Title: Mechanisms of Weight Loss in Patients Diagnosed With Achalasia
Status: Enrolling by invitation | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Vaezi, Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: 161769
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum sample will be collected for future genomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pneumatic Dilation: Subject with achalasia undergoing routine care EGD (Esophagogastroduodenoscopy) with pneumatic dilation
  Interventions: Procedure: pneumatic dilation
- Surgical Myotomy: Subject with achalasia undergoing routine care EGD with surgical myotomy
  Interventions: Procedure: surgical myotomy

INTERVENTIONS:
Procedure: pneumatic dilation — Pneumatic dilation of the lower esophageal sphincter (LES) consists of inserting a guide wire under visual control into the stomach and to pass the balloon over the guide wire. The balloon is inflated, disrupting the muscle fibers of the sphincter.
  Groups: Pneumatic Dilation
Procedure: surgical myotomy — This procedure destroys the muscles at the gastroesophageal junction, allowing the valve (LES) between the esophagus and stomach to remain open.
  Groups: Surgical Myotomy

SUMMARY:
Currently there are no existing data to determine why some achalasia patients lose weight while others do not. The purpose of this study is to gather data from patients diagnosed with achalasia to determine if differences may be identified between those who lose weight and those who do not that would help us better understand the mechanism of weight loss in this population.

DETAILED DESCRIPTION:
Patients either diagnosed with or being evaluated for achalasia and scheduled for standard clinic visits with the principal investigator as part of their routine care will be considered for participation in this study. Blood work, vital signs, and 24-hour dietary recall will be collected over a period of one year. These data will lay the foundation for future scientific endeavors to : a) assess requirements for dietary and/or nutritional supplements; b) formulate an achalasia diet; c) develop clinical practice standards; and d) design an intervention study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to provide written informed consent to participate in the study before completing any study-related procedures
2. Subject is male or female aged 18-75 years, inclusive at time of consent.
3. Subject has a documented diagnosis of achalasia based on high resolution manometry and endoscopy report.
4. Subject has been or will be scheduled to undergo either EGD with pneumatic dilation or surgical myotomy as routine care for treatment of achalasia.
5. Subject is willing and has an understanding and ability to fully comply with study procedures and restrictions defined in this protocol.

Exclusion Criteria:

1. Subject has any condition or abnormality, current or past that, in the opinion of the principal investigator, would compromise the safety of the subject or interfere with or complicate the assessment of signs or symptoms of achalasia. Such conditions may include psychiatric problems; neurologic deficits or disease; developmental delay; lung transplant; or previous gastroesophageal surgery.
2. Subject has had previous pneumatic dilation of treatment of achalasia.
3. Subject has had botulinum toxin (botox) injection for treatment of achalasia.
4. Subject has a history or high risk of noncompliance with treatment or regular clinic visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients either diagnosed with or being evaluated for achalasia and scheduled for standard clinic visits with the principal investigator or a sub-investigator as part of their routine care.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Body weight | One year
  Currently there are no existing data to determine why some achalasia patients lose weight while others do not. The purpose of this study is to determine if differences may be identified between those who lose weight and those who do not. Body weight will be monitored at study visits throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vaezi, MD,PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No